CLINICAL TRIAL: NCT01227993
Title: Extension Study for the Evaluation of Finasteride in the Treatment of Chronic Central Serous Chorioretinopathy
Acronym: CSC-Ext
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110012; 11-EI-0012
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2013-09-23 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2013-10

CONDITIONS: Retinal Disease
Keywords: Central Serous Chorioretinopathy; Finasteride; Proscar; Retinal Eye Disease
MeSH Terms: conditions — Retinal Diseases; Central Serous Chorioretinopathy | interventions — Finasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Finasteride (Experimental): Participants are treated with 5 mg oral finasteride daily when they have clinically significant subretinal fluid accumulation, defined as any subretinal fluid in the macula with a volume of at least 0.1 microliter and causing visual change such as reduced acuity, metamorphopsia, or microperimetry deficits.
  Interventions: Drug: Finasteride

INTERVENTIONS:
Drug: Finasteride
  Other Names: Proscar; Proprecia

SUMMARY:
Background:

* Central serous chorioretinopathy (CSC) is a disease in which fluid accumulates under the retina and can cause distorted vision. CSC often resolves on its own without treatment, but in chronic CSC the fluid persists and can lead to permanent visual loss. Chronic CSC may be partly caused by hormones called androgens.
* Finasteride is a drug that can modulate the effects of androgens; currently it is marketed as a treatment for male pattern baldness and benign prostate enlargement. The results of a previous brief study suggest that finasteride is safe and may help reduce the effects of chronic CSC. However, more long-term data are needed to evaluate whether finasteride is a safe and effective treatment for chronic CSC.

Objectives:

- To collect more data on the safety and effectiveness of finasteride as a treatment for chronic central serous chorioretinopathy.

Eligibility:

- Individuals who previously participated in NCT00837252 (NIH protocol 09-EI-0075), Pilot Study for the Evaluation of Finasteride in the Treatment of Chronic Central Serous Chorioretinopathy, and demonstrated clinical improvement on finasteride treatment.

Design:

* The study requires 11 visits to the NEI outpatient clinic over 5 years, with visits occurring every 6 months. Participants will be screened with a medical history, physical examination, eye examination, and blood and urine tests.
* At each visit, participants will receive a supply of finasteride pills to take every day and will need to bring any leftover finasteride pills to the following visit.
* Participants will have eye examinations to test vision, eye pressure, eye movements, and retinal thickness. Additional eye examinations will evaluate the retina's sensitivity to light and study the blood vessels and flow of blood in the eyes.
* Blood and urine samples will be taken throughout the study.
* After the end of the study, participants may be able to speak to their doctor about continuing finasteride treatments with a prescription.

DETAILED DESCRIPTION:
Objective: Central serous chorioretinopathy (CSC) is a choroidal disorder characterized by an accumulation of serous fluid under the retina. Although acute CSC tends to spontaneously resolve on its own with minimal sequelae, chronic CSC tends to persist and lead to irreversible visual loss. The pathogenesis of CSC is complex; however, systemic androgens may be involved. A recent study NCT00837252 (NIH protocol 09-EI-0075), "Pilot Study for the Evaluation of Finasteride in the Treatment of Chronic Central Serous Chorioretinopathy," suggested that finasteride, an androgen modulating medication that is widely used in the treatment of various other conditions, may be efficacious as a treatment for chronic CSC. The objective of this study is to continue evaluation of participants in the completed NCT00837252 (NIH protocol 09-EI-0075) who clinically responded to treatment with finasteride.

Study Population: Up to five participants previously enrolled in NCT00837252 (NIH protocol 09-EI-0075) who demonstrated clinical improvement on finasteride treatment.

Design: This is a 5-year pilot extension study to allow participants who demonstrated clinical improvement with finasteride for chronic CSC to continue receiving finasteride as an off-label treatment. Study visits will occur every six months over the 5-year duration. Participants will receive finasteride when they have serous fluid present, unless deemed chronic non-responders (defined as serous fluid unchanged as compared to baseline or serous fluid stabilized with no further improvement while on finasteride treatment).

Outcome Measures: The primary outcome will be the change in best-corrected visual acuity (BCVA) at two years compared to baseline. Secondary outcome measures include the annual changes in BCVA, changes in subretinal fluid volume as measured on optical coherence tomography (OCT) (a 30% reduction in subretinal fluid from baseline is considered a "treatment success" by NEI standards), changes in leakage as observed on fluorescein angiography (FA), changes in plaque size as observed on indocyanine green angiography (ICG), changes in fundus autofluorescence patterns as observed on fundus autofluorescence (FAF) imaging, changes in microperimetry patterns, changes in serum levels of testosterone and dihydrotestosterone (DHT), as well as changes in urine levels of cortisol.

ELIGIBILITY:
INCLUSION CRITERIA:

Participant previously participated in NCT00837252 (NIH protocol 09-EI-0075), Pilot Study for the Evaluation of Finasteride in the Treatment of Chronic Central Serous Chorioretinopathy, and demonstrated clinical improvement, as indicated by a reduction in subretinal fluid as measured on OCT.

Participant has subretinal fluid present in the macula that has a volume of at least 0.1 microliter causing visual change (such as reduced acuity, metamorphopsia or microperimetry deficits) and warrants treatment.

Participant must understand and sign the protocol's informed consent document.

Participant agrees to take the appropriate precautions to ensure that persons who are pregnant, nursing or of childbearing potential do not handle the finasteride tablets. [All of the NCT00837252 (NIH protocol 09-EI-0075) participants were male given the male predilection of this disease.]

EXCLUSION CRITERIA:

Participant has abnormal liver function testing (LFT) as defined by elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels that are greater than twice the respective upper limits of normal (ULN) (i.e., ALT greater than 82 U/L and/or AST greater than 68 U/L). If a participant has ALT or AST levels greater than twice the ULN, the participant can be enrolled only if cleared by hepatology.

Participant is on steroid medication (oral, topical or inhaled).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Meyerle, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gomolin JE. Choroidal neovascularization and central serous chorioretinopathy. Can J Ophthalmol. 1989 Feb;24(1):20-3. PMID 2469527
- [Background] Tewari HK, Gadia R, Kumar D, Venkatesh P, Garg SP. Sympathetic-parasympathetic activity and reactivity in central serous chorioretinopathy: a case-control study. Invest Ophthalmol Vis Sci. 2006 Aug;47(8):3474-8. doi: 10.1167/iovs.05-1246. PMID 16877418
- [Background] Spahn C, Wiek J, Burger T, Hansen L. Psychosomatic aspects in patients with central serous chorioretinopathy. Br J Ophthalmol. 2003 Jun;87(6):704-8. doi: 10.1136/bjo.87.6.704. PMID 12770965
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-EI-0012.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Finasteride
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Finasteride
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Best-corrected Visual Acuity (BCVA) in the Study Eye at Two Years Compared to Baseline
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Baseline and 2 years
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Finasteride
Number analyzed (Participants) | 3
Number analyzed (eyes) | 3
ETDRS letters | 0 (5.20)

2. Secondary Outcome: Change in Best-corrected Visual Acuity (BCVA) in the Fellow Eye at Two Years Compared to Baseline
Description: as for outcome 1
Time Frame: Baseline and 2 years
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Finasteride
Number analyzed (Participants) | 3
Number analyzed (eyes) | 3
ETDRS letters | -1.00 (5.29)

3. Secondary Outcome: Change in Best-corrected Visual Acuity (BCVA) in the Study Eye at One Year Compared to Baseline
Description: as for outcome 1
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Finasteride
Number analyzed (Participants) | 3
Number analyzed (eyes) | 3
ETDRS letters | 0 (4.58)

4. Secondary Outcome: Change in Best-corrected Visual Acuity (BCVA) in the Fellow Eye at One Year Compared to Baseline
Description: as for outcome 1
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Finasteride
Number analyzed (Participants) | 3
Number analyzed (eyes) | 3
ETDRS letters | 0.33 (4.16)

5. Secondary Outcome: Change in Serum Testosterone Levels at Two Years Compared to Baseline
Description: The concentration of testosterone in blood serum was assessed from each participant at baseline and at two years. The mean change from baseline to two years is reported here in nanograms of testosterone per decaliter of serum.
Time Frame: Baseline and 2 years
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Finasteride
Number analyzed (Participants) | 3
ng/dL | -28.67 (144.05)

6. Secondary Outcome: Change in Serum DHT Levels at Two Years Compared to Baseline
Description: The concentration of dihydrotestosterone (DHT) in blood serum was assessed from each participant at baseline and at two years. The mean change from baseline to two years is reported here in picograms of DHT per milliliter of serum.
Time Frame: Baseline and 2 years
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Finasteride
Number analyzed (Participants) | 3
pg/mL | 10.67 (44.06)

7. Secondary Outcome: Change in 24-hour Urine Cortisol Levels at Two Years Compared to Baseline
Description: The amount of cortisol found in urine was assessed from each participant at baseline and at two years. The mean change from baseline to two years is reported here in micrograms.
Time Frame: Baseline and 2 years
Measure: Mean (Standard Deviation); unit: µg
Arm/Group | Finasteride
Number analyzed (Participants) | 2
µg | 2.75 (5.16)

8. Secondary Outcome: Change in Subretinal Fluid in the Study Eye as Assessed by Optical Coherence Tomography (OCT) at Two Years Compared to Baseline
Time Frame: Baseline and 2 years
Population: Due to lack of effect in other outcome measures, at investigator's discretion, data for this outcome measure was neither collected nor analyzed. As such, zero participants have data for this outcome.
Arm/Group | Finasteride
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in Subretinal Fluid in the Fellow Eye as Assessed by Optical Coherence Tomography (OCT) at Two Years Compared to Baseline
Time Frame: Baseline and 2 years
Population: as for outcome 8
Arm/Group | Finasteride
Number analyzed (Participants) | 0

10. Secondary Outcome: Change in Area of Leakage in the Study Eye as Observed on Fluorescein Angiography (FA) Imaging at Two Years Compared to Baseline
Time Frame: Baseline and 2 years
Population: as for outcome 8
Arm/Group | Finasteride
Number analyzed (Participants) | 0

11. Secondary Outcome: Change in Area of Leakage in the Fellow Eye as Observed on Fluorescein Angiography (FA) Imaging at Two Years Compared to Baseline
Time Frame: Baseline and 2 years
Population: as for outcome 8
Arm/Group | Finasteride
Number analyzed (Participants) | 0

12. Secondary Outcome: Change in Plaque Size in the Study Eye as Observed on Indocyanine Green (ICG) Imaging at Two Years Compared to Baseline
Time Frame: Baseline and 2 years
Population: as for outcome 8
Arm/Group | Finasteride
Number analyzed (Participants) | 0

13. Secondary Outcome: Change in Plaque Size in the Fellow Eye as Observed on Indocyanine Green (ICG) Imaging at Two Years Compared to Baseline
Time Frame: Baseline and 2 years
Population: as for outcome 8
Arm/Group | Finasteride
Number analyzed (Participants) | 0

14. Secondary Outcome: Change in Autofluorescence Patterns in the Study Eye as Observed on Fundus Autofluorescence (FAF) Imaging at Two Years Compared to Baseline
Time Frame: Baseline and 2 years
Population: as for outcome 8
Arm/Group | Finasteride
Number analyzed (Participants) | 0

15. Secondary Outcome: Change in Autofluorescence Patterns in the Fellow Eye as Observed on Fundus Autofluorescence (FAF) Imaging at Two Years Compared to Baseline
Time Frame: Baseline and 2 years
Population: as for outcome 8
Arm/Group | Finasteride
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Finasteride
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finasteride (N=3)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotrasferase increased (Investigations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No